CLINICAL TRIAL: NCT01625351
Title: A Phase I Study of CD45RA+ Depleted Haploidentical Stem Cell Transplantation in Children With Relapsed or Refractory Solid Tumors and Lymphomas
Brief Title: A Study of CD45RA+ Depleted Haploidentical Stem Cell Transplantation in Children With Relapsed or Refractory Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: CURE Childhood Cancer, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RADIANT; NCI-2012-00588 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ewing Sarcoma; Gastrointestinal Tumor; Germ Cell Tumor; Hepatic Tumor; Lymphoma; Wilms Tumor; Rhabdoid Tumor; Clear Cell Carcinoma; Renal Cell Carcinoma; Melanoma; Neuroblastoma; Rhabdomyosarcoma; Non-rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Digestive System Neoplasms; Neoplasms, Germ Cell and Embryonal; Carcinoma, Hepatocellular; Lymphoma; Wilms Tumor; Rhabdoid Tumor; Adenocarcinoma, Clear Cell; Carcinoma, Renal Cell; Melanoma; Neuroblastoma; Rhabdomyosarcoma | interventions — Alemtuzumab; fludarabine; Sirolimus; Busulfan; Melphalan; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Participants to undergo transplantation. They receive alemtuzumab, fludarabine, sirolimus, busulfan, melphalan, and stem cells.
  Participants treated after activation of protocol revision 2.3 on 06/05/2014 have not and will not receive sirolimus as part of their therapy.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: alemtuzumab; Drug: fludarabine; Drug: sirolimus; Drug: Busulfan; Drug: melphalan; Biological: stem cells; Device: CliniMACS

INTERVENTIONS:
Drug: alemtuzumab — Patients receive alemtuzumab on days -14 through -12 (Day 0 = stem cell transplantation).
  Other Names: CAMPATH-1H; Campath(R)
Drug: fludarabine — Patients receive fludarabine phosphate on days -11 through -7. (Day 0 = stem cell transplantation.)
  Other Names: Fludara(R)
Drug: sirolimus — Patients receive sirolimus beginning on day -1 with taper beginning on day 90. (Day 0 = stem cell transplantation.)
  Participants treated after activation of protocol revision 2.3 on 06/05/2014 have not and will not receive sirolimus as part of their therapy.
  Other Names: Rapamycin; Rapamune(R)
Drug: Busulfan — Patients receive busulfan on days -6 through -3. (Day 0 = stem cell transplantation.)
  Other Names: Busulfex(R); Myleran(R)
Drug: melphalan — Patients receive melphalan on days -2 and -1. (Day 0 = stem cell transplantation.)
  Other Names: L-phenylalanine mustard; phenylalanine mustard; L-PAM; L-sarcolysin
Biological: stem cells — Patients undergo CD3 depleted haploidentical hematopoietic stem cell transplant (HSCT) on day 0. Patients also undergo CD45RA depleted HSCT infusion on day 1. (Day 0 = stem cell transplantation.)
  Other Names: HSCT; Stem cell transplantation
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System

SUMMARY:
This is a phase I study designed to determine the feasibility of transplantation using a novel transplant approach that employs a two-stage haploidentical cell infusion following myeloablative conditioning. This strategy, which includes selective depletion of naïve T cells, may speed immune reconstitution thereby potentially reducing the limitations of traditional haploidentical hematopoietic stem cell transplantation (HSCT) and increasing its potential therapeutic application. Additionally, the investigators intend to explore overall survival, event-free survival, hematopoietic cell recovery and engraftment as well as infection rates and complications in these patients.

DETAILED DESCRIPTION:
Twelve participants and 12 donors will be enrolled on this study. Donors will undergo seven days of hematopoietic stem cell (HSC) mobilization followed by two apheresis collections. Each apheresis collection will be processed by the CliniMACS system.

DONORS: A mobilization regimen of granulocyte colony stimulating factor (G-CSF) will be used to obtain a peripheral blood stem cell (PBSC) product from the donor. Apheresis will be performed for a minimum of two consecutive days, including one day for each cell product delivered.

STUDY PARTICIPANTS: Participants will undergo a two-stage haploidentical cell infusion following myeloablative conditioning. The first cell infusion will be a CD3-depleted product and the second infusion will be a CD45RA-depleted product.

Primary Objective:

* To determine the feasibility of haploidentical HSCT using two infusions engineered by negative selection on the Miltenyi CliniMACS system- the first by selective depletion of CD3+ cells, followed by a second depleted of CD45RA+ cells, in children with relapsed or refractory solid tumors or lymphomas.

Secondary Objectives:

* To estimate hematopoietic cell recovery and engraftment rates for the patients.
* To estimate infection rates and complications.
* To estimate the one-year overall survival (OS) and event-free survival (EFS) for the study patients.

ELIGIBILITY:
Inclusion Criteria - Transplant Recipients:

* At least 2 years of age and less than or equal to 21 years of age.
* Histologically confirmed solid tumor or lymphoma at original diagnosis:

  * Ewing Sarcoma Family of Tumors (ESFT)
  * Gastrointestinal tumors
  * Germ Cell tumors
  * Hepatic tumors (including hepatocellular carcinoma and hepatoblastoma)
  * Lymphoma (including Hodgkin and non-Hodgkin lymphoma)
  * Kidney tumors (including Wilms tumor, rhabdoid tumors, clear cell carcinoma, and renal cell carcinoma)
  * Melanoma
  * Neuroblastoma
  * Soft tissue sarcoma (including rhabdomyosarcoma and non-rhabdomyosarcoma soft tissue sarcoma)
* Malignancy has no reasonable expectation of cure with available alternative salvage therapy.
* Has a suitable human leukocyte antigen (HLA) haploidentical donor available.
* At least two weeks since receipt of any biological therapy, chemotherapy, and/or radiation therapy.
* Has recovered from all acute NCI Common Toxicity Criteria grade II-IV acute non-hematologic toxicities from prior therapy per the judgment of the PI.
* Shortening fraction greater than or equal to 25%.
* Creatinine clearance or glomerular filtration rate (GFR) greater than or equal to 50 mL/min/1.73 m2.
* Pulse oximetry greater than or equal to 92% on room air
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) less than or equal to3 times the upper limit of the institution-established normal range.
* Direct bilirubin less than or equal to 3.0 mg/dL.
* Karnofsky or Lansky performance score of greater than or equal to 50.

Exclusion Criteria - Transplant Recipients:

* Newly diagnosed patients with no prior attempt at curative therapy.
* Any primary or active central nervous system (CNS) malignancy, including metastatic disease.
* Any active or prior malignant or pre-malignant condition of the bone marrow, excluding metastasis of the primary malignancy.
* Prior allogeneic hematopoietic stem cell transplant.
* Prior autologous stem cell transplant within previous 3 months.
* Allergy to murine products or positive human anti-mouse antibody (HAMA).
* (Female only) Known pregnancy (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
* (Female only) Breast feeding.

Inclusion Criteria - Donors:

* At least 18 years of age.
* Partially HLA matched family member.
* Human immunodeficiency virus (HIV) negative.

Exclusion Criteria - Donors:

* (Female only) Known pregnancy (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
* (Female only) Breast feeding.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of haploidentical HSCT | 30 days post transplantation
  Feasibility is defined as engraftment (ANC≥ 500/mm3 for 3 consecutive tests performed on different days) evaluated before day +30.

SECONDARY OUTCOMES:
hematopoietic cell recovery and engraftment rates | 30 days post transplantation
  They will be reported and presented descriptively. Specifically, the hematopoietic cell recovery and engraftment rates will be reported with a Blyth-Still-Casella 95% confidence interval.
infection rates and complications | up to 5 years
  The proportion of patients who develop infections and complications will be estimated and a Blyth-Still-Casella 95% confidence interval will be provided.
overall survival (OS) | up to 1 year after transplantation
  Defined based on any death. The Kaplan-Meier Estimate will be provided.
event-free survival | up to 1 year after transplantation
  The Kaplan-Meier Estimate will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Brando Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols